CLINICAL TRIAL: NCT02149758
Title: EFFECT OF SELECTIVE COX-2 INHIBITOR (ETORICOXIB) ALONG WITH SCALING AND ROOT PLANING (SRP) ON CLINICAL PARAMETERS AND SALIVARY LEVEL OF SUPEROXIDE DISMUTASE IN CHRONIC GENERALIZED PERIODONTITIS A DOUBLE-BLIND, PLACEBO-CONTROLLED, DOUBLE-MASKED RANDOMIZED CONTROLLED TRIAL (RCT).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tatyasaheb Kore Dental College (Other)
Responsible Party: Principal Investigator, Dr. Sumit Sharad Shetgar, BDS (Post graduate student, Tatyasaheb Kore Dental College
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: sum2141
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Cyclooxygenase Two Inhibitors; Etoricoxib; Periodontitis; Superoxide Dismutase; Saliva
Keywords: Cyclooxygenase two inhibitors; Etoricoxib; Periodontitis; Superoxide dismutase; Saliva
MeSH Terms: conditions — Periodontitis | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etoricoxib (Experimental): Etoricoxib 60 mg once daily
  Interventions: Drug: Etoricoxib
- matching placebo (Placebo Comparator): matching placebo once daily
  Interventions: Drug: Etoricoxib

INTERVENTIONS:
Drug: Etoricoxib
  Other Names: Nucoxia; Arcoxia

SUMMARY:
The hypothesis is that Etoricoxib act as an adjuvant to SRP in alleviating periodontal inflammation by:

1. improving clinical periodontal parameters and,
2. improving the salivary SOD levels.

ELIGIBILITY:
Inclusion Criteria:Forty patients with chronic generalized periodontitis

-

Exclusion Criteria:with system illnesses, allergies, pregnancy, history of any drug intake and periodontal treatment in past 6 months.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
change from baseline in salivary SOD level | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Sumit S. Shetgar, BDS, Principal Investigator — Tatyasaheb Kore Dental College And Research Centre
Locations (1):
- Tatyasaheb kore Dental College And Research Centre, Kolhāpur, Maharashtra, India